CLINICAL TRIAL: NCT01867697
Title: Potentially Resectable Metastatic Colorectal Cancer With Wild-type KRAS and BRAF: Alternating Chemotherapy Plus Cetuximab - A Randomised Phase II Trial
Brief Title: Nordic 8 - A Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: Nordic 8
Record Dates: First submitted 2012-06-21; First posted 2013-06-04 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Oxaliplatin; Leucovorin; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biweekly cetuximab with continuously FOLFIRI (Active Comparator): Biweekly cetuximab 500 mg/m2 in combination with FOLFIRI (irinotecan 180 mg/m2 IV, leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 46 hours 5FU infusion of 2400 mg/m2 every 2 weeks)
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Folinic Acid; Drug: Calcium Carbonate
- Biweekly cetuximab with alternating FOLFIRI and mFOLFOX6 (Experimental): Biweekly cetuximab 500 mg/m2 in combination with FOLFIRI alternating with FOLFOX6 (Oxaliplatin: 85 mg/m2 IV, leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 46 hours 5FU infusion of 2400 mg/m2 every 2 weeks)
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: Folinic Acid; Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Cetuximab
Drug: Irinotecan
Drug: Oxaliplatin
  Arms: Biweekly cetuximab with alternating FOLFIRI and mFOLFOX6
Drug: Folinic Acid
Drug: Calcium Carbonate

SUMMARY:
Nordic randomized phase II trial which evaluates whether biweekly cetuximab with alternating FOLFIRI and mFOLFOX6 is more effective than biweekly cetuximab with continuously FOLFIRI in patients with potential resectable KRAS wildtype metastatic colorectal cancer.

All patients will be randomized to biweekly cetuximab 500 mg/m2 in combination with arm A) FOLFIRI (irinotecan 180 mg/m2 IV, leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 46 hours 5FU infusion of 2400 mg/m2 every 2 weeks) or arm B) FOLFIRI alternating with FOLFOX6 (Oxaliplatin: 85 mg/m2 IV, leucovorin: 400 mg/m2 IV, 5FU bolus: 400 mg/m2 IV and 46 hours 5FU infusion of 2400 mg/m2 every 2 weeks) .

Primary objective: response rate (RECIST 1.1) in patients with with potential resectable KRAS wildtype metastatic colorectal cancer.

Secondary objectives: Resection rate, PFS, OS, Quality of life, tolerability. Biomarker evaluation to measure plasma biomarkers, Tumour blocks and sequential serum and plasma will be collected to search for markers that may predict efficacy including respectability and safety.

ELIGIBILITY:
Inclusion Criteria:

Histology and stages:

* Histologically proven adenocarcinoma in the colon or rectum
* At least 1 measurable metastatic disease manifestation according to the RECIST criteria (version 1.1)
* Potentially completely resectable or potentially curable metastatic colorectal cancer as determined by the local MDT conference and that requires tumour shrinkage before resection is possible. The following definitions are indicative:

  * 4 or more liver metastases (CRLeM) without extra-hepatic disease
  * 2 or more lung metastases (CRLuM) without hepatic or extra-hepatic disease
  * 1 or more CRLeM determined as "potentially resectable" (such as because of location) by the local MDT.
  * 1 or more CRLuM determined by the local MDT as potentially resectable (such as because of location).
  * Non-resectable primary disease with resectable CRLeM or CRLuM.

KRAS and BRAF status:

- Tumour tissue (primary or metastasis) typed as wild-type KRAS AND wild-type BRAF

General conditions:

* age > 18 years
* WHO performance status ≤ 1
* expected survival > 3 months
* sufficient bone-marrow function (Hb ≥ 6.2 µmol/l/Hb > 10 g/dl ANC ≥ 1.5 x 109/l, thrombocytes ≥ 100 x 109/l)
* sufficient kidney and liver function: total bilirubin ≤ 1.5 x upper normal limit, serum creatinine ≤ 1.25 x upper normal limit, ALAT ≤ 3 x upper normal limit and ≤ 5 x upper normal limit with liver metastases
* the patient must have signed an informed declaration of consent before being registered; this must be documentable according to national guidelines

Exclusion Criteria:

Previous treatment:

* previous chemotherapy for advanced/metastatic disease
* adjuvant chemotherapy unless completed more than 6 months before registration
* previous treatment with oxaliplatin or irinotecan
* previous treatment with cetuximab or other treatment for EGFR
* History of Inflammatory Bowel disease
* Severe or uncontrolled cardiovascular disease, congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)
* Any condition that, according to the treating physician's judgement, could prevent the planned medical/surgical treatment from being carried out responsibly (such as uncontrolled active infection, known hypersensitivity or contra-indication for the planned treatment.
* Pregnant or breast-feeding women
* Patients of fertile age who do not want to use reliable contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | March 2015 (up to 3 years)

SECONDARY OUTCOMES:
Survival (Overall survival) | June 2016 (up to 5 years)
Frequency of secondary surgical resection (R0 + R1 + R2 resections) | January 2015 (up to 3 years)
Frequency of secondary micro-radical surgical resection (R0 resection) | March 2015 (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, MD, PhD, Principal Investigator — Odense University Hospital; Halfdan Sørbye, Professor, MD, Principal Investigator — Haukeland University Hospital; Bengt Glimelius, Professor, MD, Principal Investigator — Akademiske Sygehus, Uppsala University
Locations (12):
- Denmark (9):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Hospital, Esbjerg
  - Herlev University Hospital, Herlev
  - Herning Hospital, Herning
  - Naestved Hospital, Næstved
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Trondheim University Hospital, Trondheim
- Akademiska University Hospital, Uppsala, Sweden